CLINICAL TRIAL: NCT04099251
Title: A Phase 3, Randomized, Double-Blind Study of Adjuvant Immunotherapy With Nivolumab Versus Placebo After Complete Resection of Stage IIB/C Melanoma
Brief Title: Effectiveness Study of Nivolumab Compared to Placebo in Prevention of Recurrent Melanoma After Complete Resection of Stage IIB/C Melanoma
Acronym: CheckMate76K
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CA209-76K; 2019-001230-34 (EudraCT Number); U1111-1229-8927 (Other: UTN Number)
Expanded Access: NCT03126643 (Approved for marketing)
Record Dates: First submitted 2019-09-20; First posted 2019-09-23 (Actual); Results first posted 2023-07-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Nivolumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nivolumab (Experimental)
  Interventions: Biological: Nivolumab
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Nivolumab — Specified dose on specified days
  Other Names: Opdivo
  Arms: Nivolumab
Other: Placebo — Specified dose on specified days
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effectiveness of nivolumab adjuvant immunotherapy compared to placebo in adults and pediatric participants after complete resection of Stage IIB/C melanoma with no evidence of disease (NED) who are at high risk for recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Had a negative sentinel lymph node biopsy
* Participant has not been previously treated for melanoma
* ECOG 0 or 1
* Participants must have been diagnosed with histologically confirmed, Resected, Stage IIB/C cutaneous melanoma

Exclusion Criteria:

* History of ocular or mucosal melanoma.
* Pregnant or nursing women
* Participants with active known or suspected autoimmune disease
* Known history of allergy or hypersensitivity to study drug components
* Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, anti-CTLA-4 antibody, or agents that target IL-2 pathways, T-cell stimulators, or checkpoint pathways

Other protocol defined inclusion/exclusion criteria apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 790 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2027-06-29 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (130):
- United States (32):
  - Local Institution - 0088, Birmingham, Alabama
  - Local Institution - 0126, Tucson, Arizona
  - Local Institution - 0087, Springdale, Arkansas
  - Local Institution - 0080, Los Angeles, California
  - Local Institution - 0077, San Francisco, California
  - Local Institution - 0119, San Francisco, California
  - Local Institution - 0122, San Jose, California
  - Local Institution - 0121, Vallejo, California
  - Local Institution - 0109, Vallejo, California
  - Local Institution - 0120, Vallejo, California
  - Local Institution - 0091, Aurora, Colorado
  - Local Institution - 0089, Washington D.C., District of Columbia
  - Local Institution - 0141, Atlanta, Georgia
  - Local Institution - 0132, Chicago, Illinois
  - Local Institution - 0135, Baltimore, Maryland
  - Local Institution - 0078, Boston, Massachusetts
  - Local Institution - 0127, Boston, Massachusetts
  - Local Institution - 0143, Boston, Massachusetts
  - Local Institution - 0151, Minneapolis, Minnesota
  - Local Institution - 0081, Robbinsdale, Minnesota
  - Local Institution - 0079, Omaha, Nebraska
  - Local Institution - 0093, Hackensack, New Jersey
  - Local Institution - 0094, New York, New York
  - Local Institution - 0086, Charlotte, North Carolina
  - Local Institution - 0099, Cleveland, Ohio
  - Local Institution - 0076, Portland, Oregon
  - Local Institution - 0092, Allentown, Pennsylvania
  - Local Institution - 0031, Pittsburgh, Pennsylvania
  - Local Institution - 0148, Germantown, Tennessee
  - Local Institution - 0144, Austin, Texas
  - Local Institution - 0085, Dallas, Texas
  - Local Institution - 0090, Fairfax, Virginia
- Australia (12):
  - Local Institution - 0018, Waratah, New South Wales
  - Local Institution - 0025, Westmead, New South Wales
  - Local Institution - 0016, Wollstonecraft, New South Wales
  - Local Institution - 0105, Cairns, Queensland
  - Local Institution - 0017, Greenslopes, Queensland
  - Local Institution - 0024, Herston, Queensland
  - Local Institution - 0138, Southport, Queensland
  - Local Institution - 0019, Box Hill, Victoria
  - Local Institution - 0125, Geelong, Victoria
  - Local Institution - 0128, Malvern, Victoria
  - Local Institution - 0106, Melbourne, Victoria
  - Local Institution - 0104, Nedlands, Western Australia
- Austria (4):
  - Local Institution - 0049, Graz
  - Local Institution - 0051, Innsbruck
  - Local Institution - 0050, Salzburg
  - Local Institution - 0048, Vienna
- Belgium (4):
  - Local Institution - 0028, Charleroi
  - Local Institution - 0011, Ghent
  - Local Institution - 0008, Kortrijk
  - Local Institution - 0010, Liège
- Canada (8):
  - Local Institution - 0134, Calgary, Alberta
  - Local Institution - 0133, Vancouver, British Columbia
  - Local Institution - 0131, Halifax, Nova Scotia
  - Local Institution - 0142, Hamilton, Ontario
  - Local Institution - 0124, Kingston, Ontario
  - Local Institution - 0140, Toronto, Ontario
  - Local Institution - 0116, Montreal, Quebec
  - Local Institution - 0123, Sherbrooke, Quebec
- Czechia (3):
  - Local Institution - 0074, Prague, Praha 2
  - Local Institution - 0075, Ostrava-Poruba
  - Local Institution - 0073, Prague
- Denmark (3):
  - Local Institution - 0007, Aarhus N
  - Local Institution - 0012, Herlev
  - Local Institution - 0013, Odense
- Finland (3):
  - Local Institution - 0014, Helsinki, Etelä-Suomen Lääni
  - Local Institution - 0015, Tampere, Pirkanmaa
  - Local Institution - 0110, Turku
- France (10):
  - Local Institution - 0113, Brest, Finistère
  - Local Institution - 0129, Besançon
  - Local Institution - 0112, Bordeaux
  - Local Institution - 0111, Lille
  - Local Institution - 0033, Marseille
  - Local Institution - 0035, Nantes
  - Local Institution - 0130, Nice
  - Local Institution - 0036, Paris
  - Local Institution - 0032, Pierre-Bénite
  - Local Institution - 0034, Villejuif
- Germany (13):
  - Local Institution - 0056, München, Bavaria
  - Local Institution - 0072, Bonn
  - Local Institution - 0061, Buxtehude
  - Local Institution - 0098, Dresden
  - Local Institution - 0054, Essen
  - Local Institution - 0062, Gera
  - Local Institution - 0114, Göttingen
  - Local Institution - 0060, Hanover
  - Local Institution - 0055, Heidelberg
  - Local Institution - 0057, Lübeck
  - Local Institution - 0100, Mainz
  - Local Institution - 0102, Regensburg
  - Local Institution - 0058, Tübingen
- Greece (3):
  - Local Institution - 0084, Athens, Attikí
  - Local Institution - 0082, Athens
  - Local Institution - 0083, Thessaloniki
- Italy (8):
  - Local Institution - 0046, Palermo, Sicily
  - Local Institution - 0040, Bergamo
  - Local Institution - 0037, Milan
  - Local Institution - 0146, Milan
  - Local Institution - 0101, Napoli
  - Local Institution - 0039, Padua
  - Local Institution - 0145, Perugia
  - Local Institution - 0038, Siena
- Netherlands (4):
  - Local Institution - 0107, Breda
  - Local Institution - 0001, Groningen
  - Local Institution - 0030, Rotterdam
  - Local Institution - 0002, Utrecht
- Norway (3):
  - Local Institution - 0063, Bergen
  - Local Institution - 0027, Grålum
  - Local Institution - 0005, Oslo
- Poland (3):
  - Local Institution - 0103, Poznan, Greater Poland Voivodeship
  - Local Institution - 0023, Gdansk
  - Local Institution - 0022, Warsaw
- Romania (3):
  - Local Institution - 0047, Cluj-Napoca
  - Local Institution - 0020, Craiova
  - Local Institution - 0021, Sector 2
- Spain (8):
  - Local Institution - 0071, Barcelona, Barcelona [Barcelona]
  - Local Institution - 0067, A Coruña
  - Local Institution - 0065, Badalona
  - Local Institution - 0066, Madrid
  - Local Institution - 0070, Madrid
  - Local Institution - 0068, Málaga
  - Local Institution - 0064, Santander
  - Local Institution - 0069, Valencia
- Sweden (2):
  - Local Institution - 0026, Örebro
  - Local Institution - 0003, Linköping, Östergötlands Län [se-05]
- Switzerland (2):
  - Local Institution - 0053, Lausanne
  - Local Institution - 0052, Zurich
- United Kingdom (2):
  - Local Institution - 0044, Cardiff
  - Local Institution - 0095, Southampton

REFERENCES:
- [Derived] Kirkwood JM, Mohr P, Hoeller C, Grob JJ, Del Vecchio M, Lord-Bessen J, Srinivasan S, Nassar A, Campigotto F, Fairbanks H, Taylor F, Lawrance R, Long GV, Weber J. Patient-reported outcomes with adjuvant nivolumab versus placebo after complete resection of stage IIB/C melanoma in the randomized phase 3 CheckMate 76 K trial. Eur J Cancer. 2025 May 2;220:115371. doi: 10.1016/j.ejca.2025.115371. Epub 2025 Mar 19. PMID 40139004
- [Derived] Kirkwood JM, Del Vecchio M, Weber J, Hoeller C, Grob JJ, Mohr P, Loquai C, Dutriaux C, Chiarion-Sileni V, Mackiewicz J, Rutkowski P, Arenberger P, Quereux G, Meniawy TM, Ascierto PA, Menzies AM, Durani P, Lobo M, Campigotto F, Gastman B, Long GV. Adjuvant nivolumab in resected stage IIB/C melanoma: primary results from the randomized, phase 3 CheckMate 76K trial. Nat Med. 2023 Nov;29(11):2835-2843. doi: 10.1038/s41591-023-02583-2. Epub 2023 Oct 16. PMID 37845511
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT04099251.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 980 participants were screened, of which 790 participants were randomized (526 nivolumab/264 placebo) into the study and 788 received either the Nivolumab treatment (524 participants) or placebo (264 participants). 30 eligible participants (2 from the Nivolumab treatment arm and 28 from the placebo arm) received open-label Nivolumab treatment during an optional open-label phase.
Groups:
- Nivolumab: Participants received 480 mg IV Nivolumab in an approximately 30-minute infusion on Day 1 of each 4-week treatment cycle until unacceptable toxicity, recurrence/progression, withdrawal of consent, completion of 12 months of treatment from first dose of open-label study treatment, whichever occurred first.
- Placebo: Nivolumab matched placebo (0.9% Sodium Chloride for Injection/5% Dextrose for Injection) IV in a 30-minute infusion on Day 1 of each 4-week treatment cycle until unacceptable toxicity, withdrawal of consent, completion of 12 months of treatment (from first dose of study treatment), disease recurrence, or the study ends, whichever occurred first. In the event of disease recurrence, participants on the blinded nivolumab or placebo portion will be offered the option to receive open-label on-protocol nivolumab treatment. Participants received 480 mg IV Nivolumab in a 30-minute infusion on Day 1 of each 4-week treatment cycle until unacceptable toxicity, recurrence/progression, withdrawal of consent, completion of 12 months of treatment from first dose of open-label study treatment, whichever occurred first.
Period: Pre-Treatment
Arm/Group | Nivolumab | Placebo
Started (Started=randomized) | 526 | 264
Completed (Completed=treated) | 524 | 264
Not Completed | 2 | 0
Not completed — Other reasons | 1 | 0
Not completed — Participant no longer meets study criteria | 1 | 0
Period: Blinded Treatment Phase
Arm/Group | Nivolumab | Placebo
Started | 524 | 264
Completed | 257 | 158
Not Completed | 267 | 106
Not completed — Other reasons | 16 | 7
Not completed — Disease recurrence | 26 | 41
Not completed — Adverse event unrelated to study drug | 11 | 1
Not completed — Study drug toxicity | 94 | 7
Not completed — Participant no longer meets study criteria | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Death | 6 | 2
Not completed — Withdrawal by Subject | 18 | 7
Not completed — Participant request to discontinue study treatment | 29 | 0
Not completed — Ongoing treatment | 64 | 39
Not completed — Maximum clinical benefit | 1 | 2
Period: Optional Open-Label Phase Pre-Treatment
Arm/Group | Nivolumab | Placebo
Started (Started=Number of participants enrolled in the open-label phase Eligible participants received open-label Nivolumab treatment during a follow-up phase.) | 2 | 30
Completed (Completed=received treatment) | 2 | 28
Not Completed | 0 | 2
Not completed — Participant withdrew consent after re-baseline visit | 0 | 2
Period: Optional Open-Label Phase Treatment
Arm/Group | Nivolumab | Placebo
Started (Started=received optional open-label treatment) | 2 | 28
Completed | 0 | 3
Not Completed | 2 | 25
Not completed — Disease progression/recurrence | 0 | 5
Not completed — Decision by Principal Investigator | 0 | 1
Not completed — Study drug toxicity | 0 | 2
Not completed — Ongoing treatment | 2 | 17

BASELINE CHARACTERISTICS:
Groups:
- Nivolumab: Participants received 480 mg IV Nivolumab in an approximately 30-minute infusion on Day 1 of each 4-week treatment cycle until unacceptable toxicity, withdrawal of consent, completion of 12 months of treatment (from first dose of study treatment), disease recurrence, or the study ends, whichever occurred first. Participants began study treatment (Cycle 1) within 3 calendar days of randomization. Subsequent cycles were initiated within ± 3 days of the target visit date.
- Total: Total of all reporting groups
Arm/Group | Nivolumab | Placebo | Total
Number analyzed (Participants) | 526 | 264 | 790
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.9 (13.9) | 59.3 (13.6) | 59.7 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 204 | 103 | 307
  Male | 322 | 161 | 483
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 6 | 17
  Not Hispanic or Latino | 317 | 140 | 457
  Unknown or Not Reported | 198 | 118 | 316
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 515 | 262 | 777
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 8 | 1 | 9

OUTCOME MEASURES:

1. Primary Outcome: Recurrence Free Survival (RFS)
Description: Recurrence Free Survival (RFS) is defined as the time between the date of randomization and the date of first recurrence (local, regional or distant metastasis), new primary melanoma (including melanoma in situ), or death (whatever the cause), whichever occurs first. For participants who remain alive and whose disease has not recurred or did not die, RFS will be censored on the date of last evaluable disease assessment. For those participants who remained alive and had no recorded post-randomization tumor assessment, RFS will be censored on the day of randomization.
Time Frame: From randomization up to the date of first recurrence, new primary melanoma, or death (whatever the cause), whichever occurs first (up to 32 months)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab | Placebo
Number analyzed (Participants) | 526 | 264
Months | NA [28.52 to NA] — Median and upper limit not calculated due to insufficient number of events. | NA [21.62 to NA] — Median and upper limit not calculated due to insufficient number of events.
Statistical Analysis 1: Comparison: Nivolumab vs Placebo; Test type: Superiority; p < 0.0001, Regression, Cox; Hazard Ratio (HR) = 0.42, 95% CI 2-sided [0.30 to 0.59]

2. Secondary Outcome: Distant Metastasis-Free Survival (DMFS)
Description: Investigator-assessed distant metastasis-free survival (DMFS) is defined as the time between the date of randomization and the date of first distant metastasis or date of death (whatever the cause), whichever occurs first. Participants with no baseline disease assessment, no on-study disease assessments and no death, and no distant metastasis and no death will be censored. Participants with no baseline disease assessment and no on-study disease assessments and death are censored on the date of randomization. Participants with no recurrence and no death will be censored on the date of their last evaluable disease assessment.
Time Frame: From randomization up to the date of first distant metastasis or date of death (whatever the cause), whichever occurs first (up to approximately 32 months)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab | Placebo
Number analyzed (Participants) | 526 | 264
Months | NA [28.52 to NA] — Median and upper limit not calculated due to insufficient number of events. | NA [NA to NA] — Median, lower and upper limit not calculated due to insufficient number of events.

3. Secondary Outcome: Duration of Treatment on Next Line Therapy Per Investigator Assessment
Description: Duration of treatment is an investigator-assessed outcome of next-line therapy (NLT) defined as the time from first dose date of NLT to last dose date of NLT. Participants who did not stop the NLT were censored.
Time Frame: From first dose date of next-line therapy to last dose date of next-line therapy (up to approximately 32 months)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab | Placebo
Number analyzed (Participants) | 526 | 264
Months | 4.17 [2.69 to 8.38] | 11.14 [5.85 to NA] — Upper limit not calculated due to insufficient number of events

4. Secondary Outcome: Progression-Free Survival Through Next-Line Therapy
Description: Progression-free survival through next-line therapy (PFS2) is defined as the time from randomization to recurrence/objective disease progression after the start of the next-line of systemic anti-cancer therapy, or to the start of a second next-line systemic therapy, or to death from any cause, whichever occurs first. Participants who did not receive subsequent systemic anti-cancer therapy who died will be considered as having the event on the date of death. Participants who received subsequent systemic anti-cancer therapy who had a disease progression after the start of therapy will be considered as having the event on the date of disease progression. Participants who died or started second next-line therapy, the date of death or start date of second next-line therapy will be the event date, whichever is earlier. Participants who did not experience disease progression, death, or second next-line therapy will be censored on the last known alive date.
Time Frame: From randomization to recurrence/objective disease progression after the start of the next-line therapy, or to the start of a second next-line systemic therapy, or to death from any cause, whichever occurs first (up to approximately 32 months)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab | Placebo
Number analyzed (Participants) | 526 | 264
Months | NA [NA to NA] — Median, lower and upper limit not calculated due to insufficient number of events | NA [NA to NA] — Median, lower and upper limit not calculated due to insufficient number of events

5. Secondary Outcome: Number of Participants Experiencing Adverse Events (AEs)
Description: An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment. Adverse events are graded on a scale from 1 to 5, with Grade 1 being mild and asymptomatic; Grade 2 is moderate requiring minimal, local or noninvasive intervention; Grade 3 is severe or medically significant but not immediately life-threatening; Grade 4 events are usually severe enough to require hospitalization; Grade 5 events are fatal.
Time Frame: From first dose up to 30 days post last dose of the blinded phase (up to 13 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab | Placebo
Number analyzed (Participants) | 524 | 264
Participants
  Any Grade | 502 | 229
  Grade 3-4 | 115 | 32

6. Secondary Outcome: Number of Participants Experiencing Adverse Events Leading to Discontinuation
Description: An Adverse Event (AE) is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medical treatment or procedure that may or may not be considered related to the medical treatment or procedure.
Time Frame: From first dose up to 30 days post last dose of the blinded phase (up to 13 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab | Placebo
Number analyzed (Participants) | 524 | 264
Participants | 91 | 9

7. Secondary Outcome: Number of Participants Experiencing Select Adverse Events
Description: The number of participants experiencing all-cause select adverse events (AEs). An AE is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medical treatment or procedure that may or may not be considered related to the medical treatment or procedure.
Time Frame: From first dose up to 30 days post last dose of the blinded phase (up to 13 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab | Placebo
Number analyzed (Participants) | 524 | 264
Participants
  Endocrine | 116 | 14
  Gastrointestinal | 122 | 41
  Hepatic | 86 | 35
  Pulmonary | 10 | 1
  Renal | 30 | 10
  Skin | 217 | 64
  Hypersensitivity/Infusion Reactions | 33 | 2

8. Secondary Outcome: Number of Participants Experiencing Serious Adverse Events (SAEs)
Description: A Serious Adverse Events (SAE) is defined as any untoward or unfavorable medical occurrence in a participants that results in death, is life threatening, or places the participant at immediate risk of death from the event as it occurred, requires or prolongs hospitalization, causes persistent or significant disability or incapacity, results in congenital anomalies or birth defects, and is another condition which investigators judge to represent significant hazards.
Time Frame: From first dose up to 30 days post last dose of the blinded phase (up to 13 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab | Placebo
Number analyzed (Participants) | 524 | 264
Participants | 74 | 29

9. Secondary Outcome: Number of Participants Experiencing Death
Description: All study participants who died during the blinded phase of the study following treatment.
Time Frame: From first dose up to 30 days post last dose of the blinded phase (up to 13 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab | Placebo
Number analyzed (Participants) | 524 | 264
Participants | 14 | 8

10. Secondary Outcome: Number of Participants Experiencing Grade 3 or 4 Laboratory Abnormalities in Selected Hematology Parameters
Description: The number of participants experiencing Grade 3 or 4 laboratory abnormalities in the specific pre-determined hematology tests.
Time Frame: From first dose up to 30 days post last dose of the blinded phase (up to 13 months)
Population: Participants with at least one on-treatment measurement of the corresponding laboratory parameter
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab | Placebo
Number analyzed (Participants) | 512 | 261
Participants
  PLATELET COUNT | 1 | 0
  LYMPHOCYTES (ABSOLUTE), LOCAL LAB: number analyzed (Participants) | 473 | 238
  LYMPHOCYTES (ABSOLUTE), LOCAL LAB | 5 | 4
  ABSOLUTE NEUTROPHIL COUNT | 0 | 1

11. Secondary Outcome: Number of Participants Experiencing Laboratory Abnormalities in Selected Liver Parameters
Description: The number of participants experiencing laboratory abnormalities in the specific pre-determined liver tests.
Time Frame: From first dose up to 30 days post last dose of the blinded phase (up to 13 months)
Population: Participants with at least one on-treatment measurement of the corresponding laboratory parameter
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab | Placebo
Number analyzed (Participants) | 513 | 261
Participants
  ALT OR AST > 3XULN | 29 | 5
  ALT OR AST > 5XULN | 16 | 2
  ALT OR AST > 10XULN | 6 | 0
  ALT OR AST > 20XULN | 2 | 0
  TOTAL BILIRUBIN > 2XULN | 3 | 5
  ALP > 1.5XULN: number analyzed (Participants) | 512 | 261
  ALP > 1.5XULN | 20 | 1

12. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time between the date of randomization and the date of death. For those without documentation of death, OS will be censored on the last date the participant was known to be alive.
Time Frame: From randomization up to the date of death or the last date the participant was known to be alive
Reporting Status: Not Posted, anticipated posting 2028-06

ADVERSE EVENTS:
Time Frame: Participants were assessed for all-cause mortality from their randomization to primary completion, (up to approximately 32 months). SAEs and Other AEs were assessed from first dose to 100 days following last dose (up to approximately 32 months)
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication.
Groups:
- Placebo: Nivolumab matched placebo (0.9% Sodium Chloride for Injection/5% Dextrose for Injection) IV in a 30-minute infusion on Day 1 of each 4-week treatment cycle until unacceptable toxicity, withdrawal of consent, completion of 12 months of treatment (from first dose of study treatment), disease recurrence, or the study ends, whichever occurred first.
- Open-Label Nivolumab: In the event of disease recurrence, participants on the blinded nivolumab or placebo portion will be offered the option to receive open-label on-protocol nivolumab treatment. Participants received 480 mg IV Nivolumab in an approximately 30-minute infusion on Day 1 of each 4-week treatment cycle until unacceptable toxicity, recurrence/progression, withdrawal of consent, completion of 12 months of treatment from first dose of open-label study treatment, whichever occurred first.
Arm/Group | Nivolumab | Placebo | Open-Label Nivolumab
All-Cause Mortality (participants affected / at risk) | 14/526 | 8/264 | 2/32
Serious Adverse Events (participants affected / at risk) | 95/524 | 37/264 | 5/30
Other Adverse Events (participants affected / at risk) | 464/524 | 194/264 | 20/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab (N=524) | Placebo (N=264) | Open-Label Nivolumab (N=30)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 2 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0
Left ventricular failure (Cardiac disorders) | 1 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0
Myocarditis (Cardiac disorders) | 2 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 3 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 0
Hypophysitis (Endocrine disorders) | 1 | 0 | 0
Hypopituitarism (Endocrine disorders) | 2 | 0 | 0
Lymphocytic hypophysitis (Endocrine disorders) | 1 | 0 | 0
Glaucoma (Eye disorders) | 0 | 1 | 0
Uveitis (Eye disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Autoimmune colitis (Gastrointestinal disorders) | 0 | 1 | 0
Autoimmune enteropathy (Gastrointestinal disorders) | 1 | 0 | 0
Autoimmune pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 4 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 2 | 0 | 0
Volvulus (Gastrointestinal disorders) | 0 | 0 | 1
General physical health deterioration (General disorders) | 0 | 0 | 1
Generalised oedema (General disorders) | 2 | 0 | 0
Impaired healing (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Sudden death (General disorders) | 0 | 1 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 2 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0 | 0
Contrast media allergy (Immune system disorders) | 1 | 0 | 0
Abscess limb (Infections and infestations) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0
Breast cellulitis (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
COVID-19 (Infections and infestations) | 4 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 1 | 0
Diverticulitis (Infections and infestations) | 3 | 0 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 0
Herpes simplex encephalitis (Infections and infestations) | 1 | 0 | 0
Infected lymphocele (Infections and infestations) | 1 | 0 | 0
Infected seroma (Infections and infestations) | 2 | 0 | 0
Infective keratitis (Infections and infestations) | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 1
Sepsis (Infections and infestations) | 2 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tendon injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 4 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 4 | 1 | 1
Hepatic enzyme abnormal (Investigations) | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 0
Lipase increased (Investigations) | 1 | 0 | 0
Troponin increased (Investigations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Protein deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0
Steroid diabetes (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Autoimmune myositis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bone lesion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Immune-mediated myositis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Melanoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Vascular neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cerebrovascular disorder (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Embolic stroke (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Polyneuropathy (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 2 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 3 | 1 | 1
Chronic kidney disease (Renal and urinary disorders) | 1 | 0 | 0
Nephritis (Renal and urinary disorders) | 0 | 1 | 0
Nephritis allergic (Renal and urinary disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Circulatory collapse (Vascular disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
Hypertensive urgency (Vascular disorders) | 1 | 0 | 0
Lymphocele (Vascular disorders) | 1 | 0 | 0
Peripheral artery aneurysm (Vascular disorders) | 1 | 0 | 0
Vasculitis (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab (N=524) | Placebo (N=264) | Open-Label Nivolumab (N=30)
Hyperthyroidism (Endocrine disorders) | 41 | 4 | 2
Hypothyroidism (Endocrine disorders) | 63 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 22 | 14 | 1
Constipation (Gastrointestinal disorders) | 50 | 18 | 3
Diarrhoea (Gastrointestinal disorders) | 121 | 44 | 3
Dry mouth (Gastrointestinal disorders) | 41 | 10 | 4
Eructation (Gastrointestinal disorders) | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 78 | 30 | 1
Vomiting (Gastrointestinal disorders) | 19 | 12 | 2
Asthenia (General disorders) | 63 | 25 | 4
Fatigue (General disorders) | 140 | 67 | 6
Pain (General disorders) | 11 | 5 | 2
Pyrexia (General disorders) | 35 | 13 | 4
COVID-19 (Infections and infestations) | 46 | 23 | 4
Nasopharyngitis (Infections and infestations) | 15 | 7 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 28 | 2 | 0
Alanine aminotransferase increased (Investigations) | 49 | 18 | 3
Aspartate aminotransferase increased (Investigations) | 42 | 7 | 3
Blood bilirubin increased (Investigations) | 16 | 7 | 2
Blood creatine phosphokinase increased (Investigations) | 55 | 32 | 1
Lipase increased (Investigations) | 24 | 9 | 2
Decreased appetite (Metabolism and nutrition disorders) | 41 | 8 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 28 | 13 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 87 | 31 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 28 | 18 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 41 | 17 | 2
Headache (Nervous system disorders) | 65 | 34 | 1
Confusional state (Psychiatric disorders) | 2 | 1 | 2
Insomnia (Psychiatric disorders) | 16 | 15 | 0
Haematuria (Renal and urinary disorders) | 2 | 3 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 39 | 12 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 28 | 9 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 107 | 29 | 3
Rash (Skin and subcutaneous tissue disorders) | 69 | 26 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 28 | 6 | 1
Embolism (Vascular disorders) | 0 | 0 | 2
Hypertension (Vascular disorders) | 34 | 20 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-28): https://cdn.clinicaltrials.gov/large-docs/51/NCT04099251/Prot_SAP_000.pdf